CLINICAL TRIAL: NCT03598868
Title: Vortioxetine add-on Treatment Improves the Symptoms in Patients With Bipolar Depression
Acronym: ViBiD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Principal Investigator, Yong Min Ahn, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AYM-ViBiD
Record Dates: First submitted 2018-07-16; First posted 2018-07-26 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Bipolar Disorder Depression
Keywords: Bipolar Disorder; Depression, Bipolar; vortioxetine
MeSH Terms: conditions — Bipolar Disorder | interventions — Vortioxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vortioxetine (Experimental): Vortioxetine 5-20 mg
  Interventions: Drug: Vortioxetine
- Placebo (Placebo Comparator): Placebo augmentation
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vortioxetine — Augmentation : Vortioxetine 10 mg p.o. for week 1, Vortioxetine 5-20 mg p.o. for week 2,4,6.
  Other Names: Brintellix®
  Arms: Vortioxetine
Drug: Placebo — Augmentation : Placebo for week 1,2,4,6
  Arms: Placebo

SUMMARY:
The purpose of this study is to validate the efficacy of Vortioxetine augmentation in bipolar disorder patients with depressive symptoms.

DETAILED DESCRIPTION:
In this study, the investigators are going to examine the efficacy of vortioxetine augmentation in bipolar disorder patients with depressive symptoms.

The study design is a double-blinded 6-week prospective study. It would be useful for clinicians because it will provide new evidence for the effect of vortioxetine in bipolar disorder patients with depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Bipolar I Disorder, Bipolar II Disorder, Other Specified Bipolar and Related Disorder, Unspecified Bipolar and Related Disorder by Diagnostic and Statistical Manual (DSM)-V criteria.
* 18 to 65 years of age
* Patients with Montgomery-Åsberg Depression Rating Scale score ≥ 23 (moderate to severe depression), after 4 weeks or more of treatment by main medication of mood stabilizer or antipsychotics
* Patients with Young Mania Rating Scale score lower than 10, after 4 weeks or more of treatment by main medication of mood stabilizer or antipsychotics

Exclusion Criteria:

* Currently experiencing manic, hypomanic, or mixed episode
* Comorbid with serious medical illness
* Comorbid with substance use disorder, medical illness or other neurologic disorder that may have caused depressive symptoms other than by bipolar disorder
* Pregnancy or Breastfeeding women
* Those who are hypersensitive to the main or other ingredient of the medication
* Currently on Monoamine oxidase (MAO) inhibitor or those who have discontinued MAO inhibitor in the last 14 days
* Severe liver disease, severe renal disease
* Bleeding tendency/disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-08-08 (Actual); Primary Completion 2021-09-25 (Estimated); Study Completion 2021-09-25 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) | 6 weeks
  change of Montgomery-Asberg Depression Rating Scale (MADRS)

SECONDARY OUTCOMES:
Clinical Global Impressions (CGI) scale | 6 weeks
  change of Clinical Global Impressions (CGI) scale
Digit Symbol Substitution Test (DSST) | 6 weeks
  change of Digit Symbol Substitution Test (DSST)
Medication diary | 6 weeks
  compliance assessment

CONTACTS AND LOCATIONS:
Overall Officials: Yong Min Ahn, MD, PHD, Principal Investigator — Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Inha University Hospital, Incheon
  - Seoul National University Hospital, Seoul